CLINICAL TRIAL: NCT05826405
Title: Efficacy and Safety of Oral Cashew Nut Immunotherapy in Children (CAJESITO)
Acronym: CAJESITO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Amandine DIVARET-CHAUVEAU, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: FORM-03935
Record Dates: First submitted 2023-04-07; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Allergy;Food; Allergy, Nut
Keywords: allergy; food allergy; cashew nut allergy; oral immunotherapy; pistachio allergy
MeSH Terms: conditions — Food Hypersensitivity; Nut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cashew Nut allergic
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, it's an observational study

SUMMARY:
The objectives of the CAJESITO study are (i) to assess the tolerance of oral cashew nut immunotherapy, by describing the frequency and severity of allergic reactions during oral cashew nut immunotherapy and (ii )to assess the risk factors for severe allergic reactions during oral cashew nut immunotherapy (predictive factors, associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of 18 with a proven allergy to cashew nuts and followed in the pediatric allergology unit of the University Hospital of Nancy.
* Patients who have received oral cashew nut immunotherapy for at least 18 months as of 02/28/2023

Exclusion Criteria:

* Patients who have received oral cashew nut immunotherapy for less than 18 months.
* Patients lost to follow-up for more than 3 years, i.e. last consultation dating from 2020 or earlier

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients from 0 to 18 years old followed in allergology at the University Hospital of Nancy benefiting from oral immunotherapy with cashew nuts for at least 18 months as of 02/28/2023
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Number of allergic reaction | during 6 months

SECONDARY OUTCOMES:
Predictive factor of good tolerance | during 6 months
  age at onset
antibody variation | during 6 months
  Modification of level of specific IgE and IGg4 with cashew nuts
sustained unresponsiveness | 9 months
  Tolerance of 1, 2, 4, 8g in isolated doses and 15g in total cumulative dose of cashew nuts during an oral challenge test with cashew nuts 3 months after stopping the daily consumption of 2g of cashew nuts
oral tolerance of pistachio | 6 months
  Tolerance of 1, 2, 4, 8g in isolated doses and 15g in total cumulative dose of pistachio during an oral provocation test with pistachio 3 months after stopping the daily consumption of 2g of cashew nuts
Predictive factor of good tolerance | 6 months
  antecedent of severe allergic reaction
Predictive factor of good tolerance | 6 months
  initial reactogenic threshold
Predictive factor of good tolerance | 6 months
  presence atopy (asthma, food allergy or atopic dermatitis)
Predictive factor of good tolerance | 6 months
  initial specific IgE and Ana o3 levels